CLINICAL TRIAL: NCT06744166
Title: Effect of Transcutaneous Electrical Nerve Stimulation Based on Wrist-ankle Acupuncture Theory on Postoperative Pain After Video-assisted Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Jia-feng Wang, associate chief physician, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TENS-WAA-VATS
Record Dates: First submitted 2024-12-15; First posted 2024-12-20 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain; Video-assisted Thoracoscopic Surgery (VATS)
Keywords: Video-assisted thoracoscopic surgery (VATS); Postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS-WAA group (Experimental): Patients assigned to the TENS-WAA group will receive transcutaneous electrical nerve stimulation (TENS) based on Wrist-Ankle Acupuncture theory (WAA) for a duration of 30 minutes after anesthesia induction, as well as at 8 hours and 24 hours postoperatively.
  Interventions: Device: TENS-WAA
- sham TENS-WAA group (Sham Comparator): Patients assigned to the sham TENS-WAA group will receive sham stimulation （without stimulation）for a duration of 30 minutes after anesthesia induction, as well as at 8 hours and 24 hours postoperatively.
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: TENS-WAA — Patients assigned to the TENS-WAA group will receive transcutaneous electrical nerve stimulation based on Wrist-Ankle Acupuncture theory for a duration of 30 minutes after anesthesia induction, as well as at 8 hours and 24 hours postoperatively. According to the principles of WAA, two pairs of TENS-WAA (Wuxi Jiajian Medical Device Co., Ltd.) electrode pads will be placed on the upper area 2 and 3 with the skin of the treatment area exposed, and the upper and lower juxtaposition method will be adopted. Upper area 2 is at the middle of the palmar side of the forearm, between the palmaris longus and flexor carpi radialis. Upper area 3 is between the edge of the radius and the radial artery. Stimulation parameters of TENS-WAA are alternating dense-disperse wave with a frequency of 2Hz and a pulse width of 200μs, and a frequency of 100Hz with a pulse width of 150μs, alternating every 3 seconds ，intensity required to reach the maximum tolerable level without causing pain.
  Arms: TENS-WAA group
Device: Sham (No Treatment) — Patients assigned to the sham TENS-WAA group will receive sham stimulation for a duration of 30 minutes after anesthesia induction, as well as at 8 hours and 24 hours postoperatively. Researchers will attach the electrode patches at the same location, set the parameters to the same frequency, pulse width, and minimum current intensity as the TENS-WAA group, but do not activate the device, leaving it in place for 30 minutes at each time point.
  Arms: sham TENS-WAA group

SUMMARY:
At present, surgical resection remains one of the main methods for the radical treatment of lung cancer. Compared with traditional thoracotomy, Video-assisted Thoracoscopic Surgery (VATS) offers obvious advantages, such as less surgical trauma and rapid postoperative recovery. However, a certain proportion of patients will still experience moderate to severe pain after undergoing VATS. Postoperative acute pain can lead to increased postoperative pulmonary complications, prolonged hospital stays, and increased treatment costs. Additionally, it is also associated with the development of postoperative chronic pain. Therefore, effective pain management after VATS is crucial.

Researchers will compare Transcutaneous Electrical Nerve Stimulation (TENS) based on Wrist-Ankle Acupuncture theory (TENS-WAA) with a sham stimulation regimen to determine whether TENS-WAA can relieve postoperative pain in patients undergoing thoracoscopic lung resection. This study aims to enrich the existing postoperative analgesia schemes and provide a reliable basis for its clinical promotion.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* American Society of Anesthesiologists (ASA) physical status of I-III
* Patients scheduled for elective unilateral lobectomy via video-assisted thoracoscopic surgery (VATS) for lung cancer under general anesthesia
* Informed consent signed

Exclusion Criteria:

* History of liver, kidney, heart, lung, or brain disease
* Psychiatric disorder or cognitive impairment
* Chronic pain, daily use of analgesics, or alcohol dependence
* Routine or recent acupuncture treatment
* Contraindications to TENS (with pacemaker or metallic implants, allergy to surface electrodes, with skin sensory disorders, skin ulceration, unhealed scars, or adhesions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
The dynamic VAS score | at 24 hours after surgery
  Independent investigators will assess the postoperative dynamic pain (pain during activities or coughing) by utilizing a visual analogue scale (VAS) ranging from 0 to 10. The two ends of the straight line represent "no pain at all" and "the worst pain imaginable," respectively. Patients are required to mark their corresponding position on the line based on their perception of pain, and the numerical value corresponding to this position serves as the patient's pain score.

SECONDARY OUTCOMES:
The static VAS score | at 6 hours, 12 hours, 24 hours and 48 hours after surgery
  Postoperative static pain (pain at rest) will be quantified using the VAS.
The dynamic VAS score | at 6 hours, 12 hours and 48 hours after surgery
  Postoperative dynamic pain (pain during activities or coughing) will be quantified using the VAS.
Opioid consumption during surgery | at the end of the surgery
  The consumption of opioids during the surgery will be converted into morphine equivalent, and then the total will be calculated.
Postoperative opioid consumption | at 48 hours after surgery
  The consumption of opioids within 48 hours after surgery will be converted into morphine equivalent.
Consumption of NSAIDs | at 48 hours after surgery
  The consumption of Non-steroidal Anti-inflammatory Drugs within 48 hours after surgery will be recorded.
The 15-item QoR score | at 24 hours and 48 hours after surgery
  The 15-item QoR score is used to assess the quality of recovery after surgery, which ranges from 0 to 150, and higher QoR-15 scores indicate better postoperative recovery.
The HADS score | at 24 hours and 48 hours after surgery
  The Hospital Anxiety and Depression Scale (HADS) is used to evaluate patients' anxiety and depression. Scores on the HADS range from 0 to 21, and higher scores indicate more severe anxiety or depression.
The AIS score | The morning of the first day after surgery and the morning of the second day after surgery.
  The Athens Insomnia Scale (AIS) is used to assess the quality of sleep after surgery. Scores on the AIS range from 0 to 24, and higher scores indicate worse sleep quality.
Incidence of PONV | at 48 hours after surgery
  The researchers will observe whether patients experience nausea and vomiting after surgery.
The duration of hospital stay | on the 1 day of the patient's discharge from the hospital
  The period from the end of surgery to the patient's discharge from the hospital will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jiafeng Wang, M.D., Principal Investigator — Changhai hospital, Shanghai, China
Locations (1):
- Changhai hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided